CLINICAL TRIAL: NCT06300450
Title: Randomized Controlled Trial of Alert-Based Computerized Decision Support for Patients With Peripheral Artery Disease Not Prescribed Lipid-Lowering Therapy
Acronym: PAD-ALERT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Gregory Piazza, MD, MS, Associate Director, Thrombosis Research Group, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022P002171
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Artery Disease; Peripheral Vascular Diseases; Dyslipidemias
Keywords: Dyslipidemia; Peripheral Artery Disease; Peripheral Vascular Disease; Computerized Decision Support
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Dyslipidemias

STUDY DESIGN:
Intervention Model Description: 400-patient U.S.-based single-center Quality Improvement Initiative in the form of a randomized controlled trial focused on the feasibility of implementation of this patient- and provider-facing alert-based CDS (EPIC BPA)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators and outcomes assessors will be blinded to the assignment of the clinician to the computer alert or control (non-alert) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alert (Experimental): Alert-based CDS will consist of an on-screen electronic alert that will notify the clinician that the patient has an indication for LDL-C-lowering therapy but is not prescribed any. The clinician will have the opportunity to proceed to an order template through which appropriate lipid-lowering can be prescribed. The clinician could also elect to learn more about current evidence-based recommendations for LDL-C lowering in the PAD population. Finally, the clinician could elect to proceed without ordering oral LDL-C-lowering therapy or reading evidence-based recommendations for LDL-C lowering but would have to provide a rationale for not doing so.
  Interventions: Behavioral: Computer Alert
- No Alert (No Intervention): No on-screen notification will be issued to the clinician

INTERVENTIONS:
Behavioral: Computer Alert — On-screen alert-based decision support raising awareness of need for lipid-lowering therapy in patients with peripheral artery disease
  Other Names: EPIC Best Practice Advisory
  Arms: Alert

SUMMARY:
This single-center, 400-patient, randomized controlled trial assesses the impact of a patient- and provider-facing EPIC Best Practice Advisory (BPA; alert-based computerized decision support tool) to increase guideline-directed utilization of statin and statin-alternative oral LDL-C lowering therapies in patients with PAD who are not being prescribed LDL-C-lowering therapy.

DETAILED DESCRIPTION:
A Joint Task Force from the European Atherosclerosis Society and the European Society of Vascular Medicine recommends a low-density lipoprotein cholesterol (LDL-C) goal reduction of greater than 50% from baseline and a target of 55 mg/dL in patients with peripheral artery disease (PAD). An analysis of 1982 provider visits of patients with PAD in national outpatient databases in the U.S. between 2005-2012 showed that a statin was prescribed in only 33.1% of patients (Berger JS, Ladapo JA. J Am Coll Cardiol. 2017;69:2293-2300). Data from Europe demonstrates marginally better adherence to guidelines with 40% of patients with PAD prescribed a statin (Subherwal S, et al. Circulation. 2012;126:1345).

Explanations for underutilization of LDL-C-lowering therapy in patients with PAD include clinician knowledge gaps regarding evidence-based clinical practice guideline recommendations, provider inertia, the need for prior authorization for some agents, statin intolerance, and statin hesitancy. Statin intolerance is defined as the inability to tolerate a dose of statin required to sufficiently reduce cardiovascular risk and has been estimated to affect up to 15% of patients treated with statins (Banach M, et al. Arch Med Sci 2015;11:1-23 and Banach M, et al. Expert Opin Drug Saf 2015;14:935-55). While numerous statin options exist and non-statin oral options for LDL-C lowering, such as ezetimibe and bempedoic acid, are widely available, lack of awareness and inconsistent implementation contribute to underutilization in patients at high-risk for cardiovascular events, such as those with PAD. Bempedoic acid, with or without ezetimibe, is a newer option for LDL-C lowering that offers a lower prevalence of musculoskeletal side effects than statins (Diabetes Ther. 2021 Jul;12(7):1779-1789). However, familiarity with this option remains limited outside of Preventive Cardiology and Lipid Clinics.

The failure to achieve guideline-directed LDL-C targets due to clinician knowledge gaps, provider inertia, the need for prior authorization, statin intolerance, and statin hesitancy in the PAD population demonstrates similar clinical obstacles to other areas of cardiovascular medicine in which quality of care was impacted by provider and patient knowledge gaps. An alert-based computerized decision support (CDS) approach has been shown to be effective in such circumstances and could be similarly effective for optimizing lipid management in patients with PAD.

This single-center, 400-patient, randomized controlled trial assesses the impact of a patient- and provider-facing EPIC Best Practice Advisory (BPA; alert-based computerized decision support tool) to increase guideline-directed utilization of statin and statin-alternative oral LDL-C lowering therapies in patients with PAD who are not being prescribed LDL-C-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 18 years old
* Seen in Cardiovascular Medicine Clinic, Primary Care, Podiatry, Vascular Surgery, and Diabetology
* Medical history entry, visit diagnosis, or problem list entry of PAD
* Not prescribed LDL-C-lowering therapy

Exclusion Criteria:

* Patients taking a statin, ezetimibe, bempedoic acid, a PCSK9 inhibitor, inclisiran or a combination will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of prescription of oral LDL-C-lowering therapy | 90 days
  The frequency of prescription of oral LDL-C-lowering therapy will be assessed using a report from the medical record

SECONDARY OUTCOMES:
Change in LDL-C level | 6 months
  Change in LDL-C level will be assessed via the medical record

OTHER OUTCOMES:
Frequency of all-cause mortality | 6 months
  The frequency will be assessed using a report from the medical record
Frequency of major adverse cardiovascular events | 6 months
  The frequency of major adverse cardiovascular events (including myocardial infarction, stroke, hospitalization for unstable angina, or coronary revascularization) will be assessed using a report from the medical record
Frequency of major adverse limb events | 6 months
  The frequency of major adverse limb events (including amputation and peripheral artery revascularization) will be assessed using a report from the medical record
Frequency of all-cause hospitalization | 6 months
  The frequency of all-cause hospitalization will be assessed using a report from the medical record

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Piazza, Principal Investigator — BWH
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will consider IPD upon request.